CLINICAL TRIAL: NCT01011686
Title: A Phase I Clinical Study of ANT-SM (Autologous Cultured Adipose-derived Stem Cell) for the Treatment of Fecal Incontinence to Evaluate Safety
Brief Title: Safety Study of Autologous Cultured Adipose -Derived Stem Cells for the Fecal Incontinence
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Few subject enrolled
Sponsor: Anterogen Co., Ltd. (Industry)
Other Study IDs: ANT-SM-101
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

ARMS (1):
- ANT-SM (Experimental): autologous adipose-derived stem cell
  Interventions: Biological: ANT-SM

INTERVENTIONS:
Biological: ANT-SM — autologous adipose-derived stem cell

SUMMARY:
Fecal incontinence affects 18.4% adults in the community and greatly impacts quality of life. There's a problem like inconvenience, pain or allergic response in many therapeutic methods such as a surgical operation or material injection. ANT-SM is autologous adipose-derived stem cell, and so, expect of no immune responses. In this study, patients are given injection of ANT-AM in anal sphincter and followed for 4 weeks to test the safety.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Wexner's fecal incontinence score > or egal 5
* patient who has fecal incontinence for more than 6 months
* Continuity of anal sphincter at endorectal ultrasound and abnormality of anal function at anorectal manometry
* negative for urine beta-HCG for woman of childbearing age
* agreement to participate, with signed informed-consent

Exclusion Criteria:

* Anorectal surgery within the last 6 months prior to the study
* patient who is allergy to bovine-derived materials and an anesthetic
* patients with a diagnosis of auto immune disease
* Diagnosis of HBV, HCV, HIV and other infectious disease
* Patients with a diagnosis of active Tuberculosis
* Patient is pregnant or breast-feeding
* Women within 6 months post partum
* Patient who is unwilling to use an "effective" method of contraception during the study
* Patients with a diagnosis of Inflammatory Bowel Disease
* Patient who has a clinically relevant history of abuse of alcohol or drugs
* Insufficient adipose tissue for manufacturing of ANT-SM
* Patient whom investigator consider is not suitable in this study
* Patients have history of surgery for malignant cancer in the past 5 years
* Patient who has to undergo ano-rectal surgery
* Patient who has a history of artificial anal sphincter surgery
* Patient who has taken cytotoxic drugs within the last 30 days
* Patient whom investigator consider is not suitable in this study reasons for severe ano-rectal disease, severe constipation, fistula, rectal prolapsed or neurological diseases (spinal cord injury, multiple sclerosis, Parkinson's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Efficacy: Wexner's score evaluation
Safety: Clinically measured abnormality of laboratory tests and adverse events

SECONDARY OUTCOMES:
Anorectal manometry and endorectal ultrasound at week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea